CLINICAL TRIAL: NCT05586165
Title: Effects of Prompt to Bundle COVID-19 Booster and Flu Shot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey T. Fujimoto, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: covidbooster3
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; Vaccines
Keywords: COVID19; Vaccines; Text-messages; Patient Outreach; Behavioral Science; Bundling
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Holdout (No Intervention)
- Simple Reminder (Experimental)
  Interventions: Behavioral: Reminder to boost protection against COVID-19
- Flu Tag Along (Experimental)
  Interventions: Behavioral: Reminder to boost protection against COVID-19; Behavioral: Flu Tag Along
- Covid-19 Booster + Flu Bundle (Experimental)
  Interventions: Behavioral: Reminder to boost protection against COVID-19; Behavioral: COVID-19 Booster & Flu Bundle

INTERVENTIONS:
Behavioral: Reminder to boost protection against COVID-19 — Patients will receive a text message reminding them to enhance their protection against COVID-19 by getting the bivalent booster. The message will contain one link to schedule an appointment at UCLA Health and one link for scheduling an appointment at CVS Pharmacy.
  Arms: Covid-19 Booster + Flu Bundle; Flu Tag Along; Simple Reminder
Behavioral: Flu Tag Along — This message will also encourage patients to protect themselves against the flu by asking for their flu vaccine at the booster appointment (at UCLA Health) or adding the flu vaccine to the COVID-19 vaccine booster appointment (at CVS).
  Arms: Flu Tag Along
Behavioral: COVID-19 Booster & Flu Bundle — This message will simultaneously encourage patients to enhance their protection against COVID-19 and the flu and will inform them that, to save time, they can bundle two vaccines at once. Patients will learn that at UCLA Health, they can book an appointment for the booster and then ask for the flu vaccine at their appointment; at CVS Pharmacy, they can book one appointment to get both the bivalent COVID-19 booster and the flu vaccine.
  Arms: Covid-19 Booster + Flu Bundle

SUMMARY:
This randomized controlled trial investigates whether text-based reminders can increase the bivalent COVID-19 booster uptake and whether text-based reminders that mention the opportunity to bundle the COVID-19 booster with the flu shot within the same appointment can increase take-up of both the COVID-19 booster and the flu vaccine.

DETAILED DESCRIPTION:
This randomized controlled trial will test whether text-based reminders can affect the takeup of the bivalent COVID-19 booster and, in a subset of treatment, whether bundling the COVID-19 booster with the flu vaccine affects the takeup of both vaccines. The trial will be run in the Fall of 2022, and will focus on patients of UCLA Health, who have already been notified about bivalent COVID-19 boosters. This trial will include a randomly selected ~25% of patients from all UCLA Health patients eligible to receive the COVID-19 bivalent booster at the time of the study, with 35% of the remaining eligible patients randomly allocated to another trial (Pre-registration title: "Boost intentions and Facilitate Action to Promote Covid-19 Booster Take-up") and 40% randomly allocated to a third trial (Pre-registration title: "Information Provision and Consistency Framing to Increase COVID-19 Booster Uptake"). The three trials will be run simultaneously.

Patients randomly selected for this trial will be randomized at an equal share to 4 conditions: an Holdout condition that does not receive a text reminder and 3 additional conditions that receive a text message (simple reminder, Flu Tag Along, Flu and Covid-19 Bundle; see description in the Arm/Interventions section). Within each arm, patients are further randomized into one of the 33 time slots for when they will receive the text message (i.e., 3 time points per day including 9am, 12pm, 4pm for 11 days). Days 1-4 and 8-11 have slightly fewer patients than Days 5-7.

To test whether the text reminders increase booster uptake, the investigators will compare the holdout condition to the combination of the 3 reminder arms.

The investigators will address additional research questions:

1. The investigators will investigate whether reminders that mention the flu vaccine are effective at increasing booster take-up rates. For this question, the investigators will first compare booster uptake and link click rates between the two reminders that mention the flu vaccine to each other. If one reminder outperforms the other in a given outcome, the investigators will then compare the more effective of the two reminders to a) the holdout and b) the simple reminder that does not mention the flu vaccine for that given outcome. If the two reminders that mention the flu vaccine are not significantly different, the investigators will compare the average of these two reminders to a) the holdout and b) the simple reminder. The investigators will also compare the simple reminder to the holdout. For these analyses, the investigators will not only examine all patients that satisfy the inclusion/exclusion criteria but also examine just the subset of patients who have not received the flu shot in the 2022-2023 flu season or made a flu shot appointment at UCLA Health by the time of receiving the text message. Further, among the latter subset of patients, the investigators will also explore whether the reminders that mention the flu vaccine increase flu vaccine uptake, relative to the simple reminder and holdout.
2. The investigators will also explore how the effects of text reminders encouraging people to get vaccinated at UCLA/CVS vary by the scope and horizon of booster uptake measure. For this purpose, the investigators will compare the combination of the three reminders, which contain links to UCLA/CVS, with the holdout, and the investigators will analyze both booster uptake at UCLA/CVS and booster uptake in California and both at 2 weeks and 4 weeks. The investigators will do the same analyses for the additive effect of encouraging people to get flu vaccine and COVID-19 booster at the same time.
3. The investigators will explore the role of the time when a text message is sent. The investigators will examine how the effect of text reminders (i.e., the combination of the 3 reminder arms vs. holdout) varies across days and times. As additional specifications, the investigators will control for the time trend and analyze all patients who have not gotten the bivalent booster in California or scheduled a booster appointment at UCLA Health the day before the trial starts.

Analysis:

The investigators will run ordinary least squares regressions (OLS) with robust standard errors to predict the aforementioned outcome variables, except that the investigators will use a Cox proportional hazards model with administrative censoring to predict time of obtaining the booster. The significance level will be 0.05. Our regressions will include the following control variables:

* Indicators for one of the 33 time slots
* Participant age (If there will be a missing value, the investigators will replace with the mean and add a dummy variable to indicate patients with missing age)
* Indicators for participant race/ethnicity (Black non-Hispanic, Hispanic, Asian non-Hispanic, white non-Hispanic, other/mixed, unknown)
* Indicators for participant gender (male, female, other/unknown)

The investigators will test whether the main effect of sending text reminders (i.e., the combination of the 3 reminder arms vs. holdout) is robust regardless of:

* Whether the patient is female or male
* Whether the patient is white non-hispanic or racial/ethnical minority
* Whether the patient is 65+ (including 65) or below 65

The investigators will investigate the following moderators for (1) the main effect of sending text reminders and (2) the effect of encouraging people to get flu vaccine and COVID-19 booster at the same time:

* Timing of the first dose of the COVID-19 vaccine primary series
* Whether patients got at least one original booster
* Whether or not the patient received a flu shot in either the 2020-2021 season or the 2021-2022 flu season according to the patient's medical record
* How strongly the patient's neighborhood is in favor of the Republican (vs. Democratic) Party if UCLA Health eventually agrees to provide de-identified addresses (e.g., zip code) and if our sample includes patients living in Republican-leaning counties.

Additional information: Three days into this trial, the investigators learned that the supply of boosters at UCLA Health is very limited and patients could not find appointments at UCLA Health. The investigators verified that local pharmacies continue to have appointments available. Thus, the investigators updated all text messages to (1) explain that UCLA Health has limited booster appointments available, (2) no longer provide a direct link to schedule appointments at UCLA Health, and (3) instead encourage patients to make an appointment at either CVS Pharmacy or local pharmacies (depending on the arm). As a result, instead of analyzing the originally preregistered outcome measures of "booster take-up at UCLA/CVS in 2 weeks", "booster take-up at UCLA/CVS in 4 weeks", "flu vaccine take-up at UCLA/CVS in 2 weeks" and "flu vaccine take-up at UCLA/CVS in 4 weeks",the investigators will measure vaccine uptake at CVS in 2 weeks and 4 weeks. In terms of the outcome measure of "Link click rate in 1 week", the investigators will still look at whether patients click on any link in the text message.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above
* Have a mobile phone number or SMS-capable phone number in UCLA Health's database
* Having completed a COVID-19 vaccine primary series based on CAIR data
* Last COVID-19 vaccine shot (including booster shot) occurred at least two months before the date when patient list are pulled in preparation for the trial, based on CAIR data. The last two criteria meant to identify patients who are eligible for the updated booster.

Exclusion Criteria:

* Patients who have received the bivalent booster anywhere (based on CAIR data) before the day they receive the text message
* Patients who have already scheduled appointments at UCLA Health for getting the bivalent booster before the day they receive the text message

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109493 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
booster take-up at UCLA/CVS in 2 weeks | 2 weeks after getting the text message
  Whether people receive the bivalent booster at either UCLA Health or CVS Pharmacy
booster take-up at UCLA/CVS in 4 weeks | 4 week after getting the text message
  Whether people receive the bivalent booster at either UCLA Health or CVS Pharmacy

SECONDARY OUTCOMES:
Link click rate in 1 week | 1 week after getting the text message
  Whether people click on at least one link provided in the text message
booster take-up in 2 weeks | 2 weeks after getting the text message
  Whether people receive the bivalent booster at any location reporting to the California Immunization Registry (CAIR)
booster take-up in 4 weeks | 4 weeks after getting the text message
  Whether people receive the bivalent booster at any location reporting to the California Immunization Registry (CAIR)
Flu vaccine take-up at UCLA/CVS in 2 weeks | 2 weeks after getting the text message
  Whether people receive the flu vaccine at either UCLA Health or CVS Pharmacy
Flu vaccine take-up at UCLA/CVS in 4 weeks | 4 weeks after getting the text message
  Whether people receive the flu vaccine at either UCLA Health or CVS Pharmacy
Flu vaccine take-up in 2 weeks | 2 week after getting the text message
  Whether people receive the flu vaccine at at any location reporting to the California Immunization Registry (CAIR)
Flu vaccine take-up in 4 weeks | 4 weeks after getting the text message
  Whether people receive the flu vaccine at any location reporting to the California Immunization Registry (CAIR)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No